CLINICAL TRIAL: NCT02768545
Title: Pilot Study of Ezetimibe for Chronic Hepatitis C Virus (HCV) Infection in Liver Transplant Candidates (EZE-2)
Brief Title: Study of Ezetimibe for Chronic Hepatitis C Virus (HCV) Infection in Liver Transplant Candidates (EZE-2)
Acronym: EZE-2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Alejandro Soza, MD, Associate Professor, Pontificia Universidad Catolica de Chile
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-199b
Record Dates: First submitted 2016-05-08; First posted 2016-05-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Ezetimibe; Cholesterol; Enterohepatic Circulation; Bile; Feces
MeSH Terms: conditions — Hepatitis C | interventions — Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Liver transplant candidates (Experimental): Ezetimibe in a dose of 10 mg/d for 12 weeks.
  Interventions: Drug: Ezetimibe

INTERVENTIONS:
Drug: Ezetimibe — Ezetimibe 10 mg per day before and after transplant

SUMMARY:
NPC1L1 is a key transporter in the enterohepatic cycle of cholesterol. Initial in vitro and in vivo data show that blocking this receptor with ezetimibe results in delaying infection in these models. The investigators hypothesize that HCV has an enterohepatic cycle, being secreted in bile and reabsorbed either in the canalicular membrane or in the intestine by association with NPC1L1, following a path similar to the cycle of cholesterol in humans. To prove this hypothesis the investigators propose to assess the effect of ezetimibe treatment in HCV infected individuals undergoing liver transplantation to avoid or delay HCV infection. For this purpose, the investigators propose to administrate ezetimibe 10 mg/d for 12 weeks to 12 patients with chronic hepatitis C infection listed for a liver transplantation.

DETAILED DESCRIPTION:
Infection by hepatitis C virus (HCV) affects more than 170 million people in the World and 80.000 in Chile. It causes more deaths than HIV infection in the US and is a leading cause of liver transplantation in Chile. Even though treatments are evolving with new direct antiviral agents (DAAs) with increasing response rates, there are several issues with these new approaches, including toxicity, need for using interferon and ribavirin, complex algorithms of treatment, high cost, limited effectivity in certain groups (liver transplant patients) and drug interactions. Treatments targeted at host factors required for the viral cycle are becoming increasingly explored as an alternative or complement to DAAs. HCV has a very intimate connection with host lipidic pathways, altering the lipid profile, circulating bound to lipoproteins and using cholesterol receptors and intracellular mechanisms of fat metabolism. It has been recently described that NPC1L1 (Niemann-Pick C1-like 1), the intestinal receptor of cholesterol, serves as an entry factor for HCV. Interestingly, this receptor is not only expressed in the enterocytes (absorbing both endogenous and dietary cholesterol), but also in the canalicular membrane of the hepatocyte, where it functions absorbing cholesterol secreted into the canalicular lumen. NPC1L1 is, therefore, a key transporter in the enterohepatic cycle of cholesterol. Initial in-vitro and in-vivo data show that blocking this receptor with ezetimibe results in delaying infection in these models. Moreover, it has reported the case of a patient that after 3 unsuccessful treatment attempts, cleared HCV RNA with ezetimibe treatment, being the first report of the effect of ezetimibe in humans. In view of these observations, the investigators hypothesize that HCV has an enterohepatic cycle, being secreted in bile and reabsorbed either in the canalicular membrane or in the intestine by association with NPC1L1, following a path similar to the cycle of cholesterol in humans.

This possibility is further supported by the observation that HCV RNA has been detected in bile and feces of infected humans. To prove this hypothesis, the investigators propose to assess the effect of ezetimibe treatment in HCV-infected individuals. Ezetimibe is an approved and generally safe drug used for the management of hypercholesterolemia. HCV RNA and core antigen in plasma and feces will be assessed. An increase in bile or fecal HCV load after antagonizing NPC1L1 with ezetimibe will support the notion that HCV is reabsorbed in the canalicular membrane or at the intestinal level. The second part of the proposed study will be conducted in 12 patients who have chronic hepatitis C and are listed for a liver transplantation. Graft reinfection after liver transplant is universal. Here the investigators anticipate that the use of ezetimibe will directly impact on the reinfection time of the graft, by delaying or even preventing liver reinfection in some patients. Should this study be successful it will for sure have enormous implications for the design of novel management strategies for liver transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C defined as detectable HCV RNA for more than 6 months.
* Age > 18 years old.
* No current HCV antiviral treatment.
* No medications for dyslipidemia in the preceding 2 months.
* Listed in the national waiting list for liver transplant with an estimated time to transplantation of 3 months or less, either for complications of cirrhosis or for hepatocellular carcinoma.
* No abdominal surgery that could alter biliary or intestinal anatomy.
* HCV RNA level > 10.000 IU/mL.
* No evidence of sitosterolemia.
* Negative pregnancy test in urine (for females).
* Signed informed consent document.

Exclusion Criteria:

* Hepatitis B or HIV co-infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Controlled viral load | 4 weeks after liver transplantation
  Proportion of patients with HCV viral load lower than pre-transplant viral load measured at 4 weeks after liver transplant.

SECONDARY OUTCOMES:
Sustained virologic response | 12 weeks
  Percentage of participants with HCV viral load < 25 IU/mL after 12 weeks of completing treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Soza, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Departamento de Gastroenterología, Pontificia Universidad Católica de Chile, Santiago, RM, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agnello V, Abel G, Elfahal M, Knight GB, Zhang QX. Hepatitis C virus and other flaviviridae viruses enter cells via low density lipoprotein receptor. Proc Natl Acad Sci U S A. 1999 Oct 26;96(22):12766-71. doi: 10.1073/pnas.96.22.12766. PMID 10535997
- [Background] Allain CC, Poon LS, Chan CS, Richmond W, Fu PC. Enzymatic determination of total serum cholesterol. Clin Chem. 1974 Apr;20(4):470-5. No abstract available. PMID 4818200
- [Background] Beld M, Sentjens R, Rebers S, Weel J, Wertheim-van Dillen P, Sol C, Boom R. Detection and quantitation of hepatitis C virus RNA in feces of chronically infected individuals. J Clin Microbiol. 2000 Sep;38(9):3442-4. doi: 10.1128/JCM.38.9.3442-3444.2000. PMID 10970398
- [Background] Ge L, Wang J, Qi W, Miao HH, Cao J, Qu YX, Li BL, Song BL. The cholesterol absorption inhibitor ezetimibe acts by blocking the sterol-induced internalization of NPC1L1. Cell Metab. 2008 Jun;7(6):508-19. doi: 10.1016/j.cmet.2008.04.001. PMID 18522832
- [Background] Haruna Y, Kanda T, Honda M, Takao T, Hayashi N. Detection of hepatitis C virus in the bile and bile duct epithelial cells of hepatitis C virus-infected patients. Hepatology. 2001 Apr;33(4):977-80. doi: 10.1053/jhep.2001.23435. PMID 11283863
- [Background] Jia L, Betters JL, Yu L. Niemann-pick C1-like 1 (NPC1L1) protein in intestinal and hepatic cholesterol transport. Annu Rev Physiol. 2011;73:239-59. doi: 10.1146/annurev-physiol-012110-142233. PMID 20809793
- [Background] Nielsen SU, Bassendine MF, Burt AD, Martin C, Pumeechockchai W, Toms GL. Association between hepatitis C virus and very-low-density lipoprotein (VLDL)/LDL analyzed in iodixanol density gradients. J Virol. 2006 Mar;80(5):2418-28. doi: 10.1128/JVI.80.5.2418-2428.2006. PMID 16474148
- [Background] Sainz B Jr, Barretto N, Martin DN, Hiraga N, Imamura M, Hussain S, Marsh KA, Yu X, Chayama K, Alrefai WA, Uprichard SL. Identification of the Niemann-Pick C1-like 1 cholesterol absorption receptor as a new hepatitis C virus entry factor. Nat Med. 2012 Jan 8;18(2):281-5. doi: 10.1038/nm.2581. PMID 22231557
- [Background] Temel RE, Tang W, Ma Y, Rudel LL, Willingham MC, Ioannou YA, Davies JP, Nilsson LM, Yu L. Hepatic Niemann-Pick C1-like 1 regulates biliary cholesterol concentration and is a target of ezetimibe. J Clin Invest. 2007 Jul;117(7):1968-78. doi: 10.1172/JCI30060. PMID 17571164